CLINICAL TRIAL: NCT04271579
Title: Early Prostate Cancer Recurrence With PSMA PET Positive Unilateral Pelvic Lesion(s): is One-sided Salvage Extended Lymph Node Dissection Enough
Brief Title: Early Prostate Cancer Recurrence With PSMA PET Positive Unilateral Pelvic Lesion(s)
Acronym: ProsTone
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Martini-Klinik am UKE GmbH (Other)
Collaborators: University Medical Center Hamburg-Eppendorf (UKE) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ProsTone-MK-2020; DRKS00020130 (Other: German Clinical Trail Register)
Record Dates: First submitted 2020-02-12; First posted 2020-02-17 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer
Keywords: prostate cancer recurrence; salvage lymph node dissection
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Unilateral lymphnode dissection (Active Comparator): Salvage lymphnode dissection is performed on the PSMA PET positive side, according to template (obturator, iliac external, iliac internal, iliac commun) and possibly including other anatomical pelvic regions
  Interventions: Procedure: Salvage Lymphnode dissection
- bilateral Lymphnode dissection (Active Comparator): In addition, a salvage lymphnode dissection is performed on the opposite side with resection of the corresponding fields, which were taken on the PSMA-PET positive side
  Interventions: Procedure: Salvage Lymphnode dissection

INTERVENTIONS:
Procedure: Salvage Lymphnode dissection — A salvage lymphnode dissection is performed in all study patients (both arms)using standard surgical techniques (openly or DaVinci).In patients who were randomized to the bilateral pelvic lymphnode dissection group, a salvage lymphadenectomy was also performed on the opposite side with resection of the corresponding fields that were removed on the PSMA-PET positive side (th "Blinding" must be guaranteed during pathological assessment)

SUMMARY:
Significant advances in molecular nuclear medicine imaging in prostate cancer have been achieved in recent years. In particular, the introduction of prostate-specific membrane antigen (PSMA) -based tracers has significantly influenced diagnostic imaging of prostate. If cancer recurs after surgical removal of the prostate, targeted PSMA PET (positron emission tomography) can detect metastases even at very low PSA (prostate-specific Antigen) values. This increasingly allows individualized specific therapy of patients with prostate cancer recurrence. PSMA PET has now been included in national and international guidelines for the diagnosis of patients with biochemical recurrence of prostate cancer.

Especially in patients in good general condition, with potentially longer life expectancy and early localized PSA recurrence, advances in molecular imaging are increasingly turning local therapy concepts into focus. Here both, radiotherapeutic (salvage radiotherapy of the lymphatic drainage) and surgical interventions (salvage lymph node dissection = removal of the pelvic lymph nodes) are offered on an individual basis.

These regional therapies mainly aim to achieve a delay of further progression of the prostate cancer disease, and thus delay the initiation of palliative, sustained drug therapy. Previous standard or common practice at salvage lymph node dissection is the removal on both sides of the pelvic lymph nodes even if only one-sided suspicious lymph nodes are detected on imaging. Although the complications of salvage lymph node dissection are usually minor and manageable, they can still lead to impaired lymphatic drainage, leg edema, lymphocele formation or other surgical complications.

The aim of the present study is to investigate whether a unilateral pelvic lymph node dissection on the side of conspicuous PSMA PET is sufficient and a dissection on the contralateral side can be dispensed without negatively impacting oncological outcomes and thereby sparing the patient the potential additional complications of a bilateral pelvic lymph node dissection.

DETAILED DESCRIPTION:
In this prospective randomized study, patients with early biochemical recurrence after radical prostatectomy and with PSMA-PET positive unilateral pelvic metastatic lesions are assessed as to whether unilateral and bilateral salvage lymph node dissection are oncologically equivalent. For this, the following endpoints will be evaluated:

* complete biochemical response (cBR: PSA <0.2ng /ml) after salvage lymph node dissection
* biochemical freedom from recurrence without further prostate-cancer-specific therapy (time from salvage lymph node dissection to first PSA value> 0.2ng / ml)
* prostate cancer-specific therapy-free time (time from salvage lymph node dissection to initiation of prostate cancer specific therapy) In addition, the diagnostic accuracy of the preoperative PSMA PET, which led to the indication of salvage lymph node dissection, is to be investigated in the context of the study and the standardized one- or two-sided template lymph node dissection. Furthermore, it should be investigated whether there is a reduction of surgery-associated side effects in patients undergoing unilateral salvage lymph node dissection. In addition, quality of life and psychological stress of patients is systematically recorded by means of validated questionnaires. Since salvage lymph node dissection may also be carried out with the help of currently experimental preoperative labeling with PSMA ligands for easier intraoperative localization (PSMA radioguided surgery), a comparison of conventional salvage surgery and the PSMA radioguided surgery is also planned. However, if applied to patients, PSMA radioguided surgery is performed outside of the study protocol and is explicitly not part of the study protocol.

In case there is no complete biochemical response (cBR, PSA <0.2ng / ml) or, after reaching cBR, a further increase in PSA above 0.2ng / ml threshold is observed after salvage lymph node dissection, an attempt should be made to localize recurrence disease using PSMA PET. This should provide indirect information as to whether re-irradiation following salvage lymph node dissection could be a useful approach and should be investigated in future studies. However, PSMA PET is recommended in the study, but is optional and therefore to be performed outside of the study protocol.

Amendment01, Addition to the two-step consent process: First, suitable patients will be offered participation in this prospective study. If the patients consent, randomization will be carried out and the patient will be informed of the result of the randomization (unilateral or bilateral procedure). Patients will then be asked whether they would like to be treated in accordance with the randomization result. If they consent, they will be treated analogously and included in the study cohort. If they do not consent to be treated analogously to the randomization result, they will be treated as part of a study-associated control group and further observed.

ELIGIBILITY:
Inclusion Criteria:

* Patients in good general condition with life expectancy> 10 years
* Hormone-sensitive prostate cancer recurrence after radical prostatectomy (patients with status post salvage prostatectomy may be included; salvage radiotherapy for prostate fossa and / or pelvic lymph drainage after radical prostatectomy is not an exclusion criterion)
* Unilateral detection of ≤ 3 PSMA PET positive lymph node metastases in the pelvis (up ot origin of the inferior mesenteric artery)
* PSA at the time of PSMA PET imaging <4 ng / ml

Exclusion Criteria:

* Contraindication for surgery or bilateral salvage lymph node dissection
* Suspected prostate cancer recurrence in the prostate fossa (local recurrence) or extrapelvic metastasis on PSMA PET imaging
* Date of PSMA PET examination > 4 months prior to salvage lymph node dissection
* Hormone therapy within 6 months prior to study enrollment

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 397 (Estimated)
Dates: Start 2019-10-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of complete biochemical response | 24 months
  cBR: PSA <0.2ng / ml after salvage lymph node dissection without adjuvant prostate cancer specific therapy

SECONDARY OUTCOMES:
Prostate cancer-specific therapy-free survival | 12 months
  e.g. medicinal, radiotherapy, operative

CONTACTS AND LOCATIONS:
Locations (1):
- Martini-Klinik am UKE GmbH, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No